CLINICAL TRIAL: NCT00796042
Title: Interdisciplinary Pressure Management & Mobility Program as an Alternative to Bed Rest: A Pilot Study
Brief Title: Interdisciplinary Pressure Management & Mobility Program as an Alternative to Usual Care: A Pilot Study
Acronym: WOUND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Ontario Neurotrauma Foundation (Other)
Responsible Party: Principal Investigator, Dianne Bryant, Associate Professor, University of Western Ontario, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONF-2004-SCI-SC-01; ONF-2004-SCI-SC-01; NCT00569205 (obsolete NCT alias)
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Pressure Ulcer
Keywords: Pressure Ulcer; Bed Sores; Bedsore; Decubitus Ulcer; Pressure Sore; Best rest; mobility; pressure management
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Usual Care
  Interventions: Other: Usual care
- 2 (Experimental): Individualized, Community-based, Pressure management and Mobility program:
  Interventions: Other: Pressure management and Mobility program

INTERVENTIONS:
Other: Usual care — Subjects will be encouraged to implement the standard wound care protocol that is consistent with the National (CAWC) and Provincial (RNAO) best practice guidelines for the treatment of pressures ulcers. This wound care program will be customized to subject's needs based on the results of the assessment performed by the wound care specialist. A registered dietitian will review blood values associated with nutritional status and make recommendations for dietary changes. Wherever possible, implementation of this wound care program will be coordinated with the subjects' current health care team and appropriate referrals to home care agencies or specialists will be initiated where needed. Subjects assigned to this group will continue their current level of activity (bed rest). Any equipment or services will be obtained through the usual provider agencies.
  Arms: 1
Other: Pressure management and Mobility program — Subjects are provided with the same customized wound care program as the usual care group and a pressure management and mobility program that is customized to the individual's needs. This program is based on an in depth home assessment performed by a registered Occupational (OT) or Physical Therapist (PT). Pressure Management Program: A qualified OT or PT will examine the subject on all in-use surfaces and observe all transfers to identify sources of friction and shear, and any strength or balance deficits, identifying what equipment/services are required to manage pressure, improve mobility, and reduce friction and shear. Mobility Program: A qualified PT will assess strength, balance, range of motion, and functional independence with transfers and other ADLs and will develop a mobility program to optimize functional independence and improve strength and balance required for safe and effective transfers. Program to be implemented within one month of this evaluation.
  Arms: 2

SUMMARY:
People with spinal cord injuries posses many factors that increase their risk of developing pressure ulcers. Not surprisingly, approximately 82% of persons with spinal cord injury (SCI) will experience a pressure ulcer at sometime during their life. Earlier guidelines for the assessment and treatment of pressure ulcers produced by RNAO in 20027 recommended that "a client who has a pressure ulcer on a seating surface should avoid sitting." Unfortunately, this recommendation has fueled the long standing view that people with pressure ulcers should stop using their wheelchairs and return to bed. The strength of evidence assigned for this recommendation was Level=C reflecting the paucity of research evidence to support this common practice. Not only do the benefits of bed rest on healing remain to be demonstrated, there is mounting evidence that bed rest can be harmful to a person's overall health and well being. Bed rest has been shown to be strongly associated with complications in most body systems including respiratory, cardiovascular, musculoskeletal, cerebrovascular, gastrointestinal, and genital-urinary. Psychosocial complications and cognitive impacts are also well documented. Without evidence to dispel the myth that "bed rest is best" it will be difficult to change practice and avoid many of the secondary complications. This study is a pilot study to 1) determine whether pressure ulcers heal faster in individuals with SCI who receive an individualized community-based, pressure management and mobility program compared to a similar group assigned to usual care (bed rest), 2) determine the strength of the association between the intervention (pressure/mobility or bedrest) and wound healing, motor performance/independence and quality of life while adjusting for motivation to regain independence, degree of caregiver burden, and compliance with the intervention, 3) determine whether individuals with SCI who participate in a pressure/mobility management program experience fewer secondary complications than those who do not participate, 4) determine the cost-effectiveness of providing a time-efficient, pressure management and mobility program compared to bed rest.

DETAILED DESCRIPTION:
Hypothesis: Individuals with SCI who have pressure ulcers who receive an individualized, community-based, pressure management and mobility program will have better outcomes compared to a similar group of individuals who remain on bed rest (usual care).

Specific Objectives

1. To determine whether pressure ulcers heal faster in individuals with SCI who receive an individualized community-based, pressure management and mobility program compared to a similar group assigned to usual care (bed rest).
2. To determine the strength of the association between the intervention (pressure/mobility or bedrest) and wound healing, motor performance/independence and quality of life while adjusting for motivation to regain independence, degree of caregiver burden, and compliance with the intervention.
3. To determine whether individuals with SCI who participate in a pressure/mobility management program experience fewer secondary complications than those who do not participate
4. To determine the cost-effectiveness of providing a time-efficient, pressure management and mobility program compared to bed rest.
5. To formally evaluate our ability to successfully recruit eligible patients into the full study.
6. To determine the barriers and facilitators to successful implementation of a pressure management and mobility program from the perspective of the client, caregiver, and health care provider.
7. To use our experiences individualizing pressure management and mobility programs to develop a preceptorship/mentorship training program for community-based pressure/mobility management that can be transferred to other regions in Ontario through distance education.

Study Design: This pilot study is a double-blind, parallel group, randomized controlled cross-over design that will be conducted in two centres over a 1.5 year period. Rigorous pilot data will ensure that our intervention has sufficient potential to warrant further investigation, will determine whether our protocol is feasible. As such, the methods and data collection strategies laid out in this protocol are meant to mimic the full trial.

Sample population We will enroll twenty individuals with SCI living in each of the two sites (Toronto (n=10) and London (n=10)) who have a Stage II to IV pressure ulcer(s) and meet the eligibility criteria.

Screening assessment: A research assistant will contact volunteers who consent to participate in the study and assess the subject's willingness to undergo a medical and wound assessment to determine study eligibility. She/he will collect, information on SCI injury, demographics, current level of activity, wheelchair use, and wound history. This will entail a phone interview and home assessment and the research assistant will schedule the clinic visit to assess eligibility. For subjects who are interested in learning more about the study, the research assistant will schedule the clinic visit to assess eligibility.

Wound Assessment: We will arrange transportation to the wound management centre where the subject's eligibility for study participation (see Inclusion/Exclusion criteria) will be determined. The subject's current medical status and pressure sore(s) will be assessed by research personnel including a qualified wound care specialist and she/he will record detailed wound history, determine wound extent and severity, and assess the likelihood that the wound will heal over the 8 month study period. As part of this medical screen, a blood sample will be drawn and wound swab will be obtained and analyzed for key determinants of healing (metabolic disorders, anemia, nutritional deficiencies, infection). From this assessment, we will develop a treatment plan to optimize wound environment, provide nutritional supplementation, and modify factors interfering with healing.

Assignment of subjects to study groups: Following wound assessment, we will randomize ten eligible subjects from each study centre (London and Toronto) who meet eligibility criteria using the Zelen method whereby randomization to treatment group occurs prior to subject consent for participation. Those subjects allocated to intervention group will be asked to consent to participation in a randomized trial comparing usual care to a pressure management and mobility program. They will be informed that they have been randomized to receive the pressure management and mobility program. Those subjects allocated to usual care will be asked to consent to participate in a long-term prospective natural history study to document the effects of bed rest in individuals who have SCI and pressure wounds. This method of randomization reduces the considerable risk of producing a biased estimate of the effect of treatment since patients assigned to usual care are likely to feel that other study participants are receiving better care (despite the lack of evidence to support this notion). This method of blinding the patient is especially important in trials with subjective and self-report outcome measures.

Using data obtained from the assessment at the wound centre, the randomization scheme will be stratified according to two key determinants of healing; wound severity (Stage of pressure ulcer II, III, IV); 2) and the presence or absence of 2 or more abnormal blood values to ensure that the potential confounding affect on wound healing is equally dispersed between treatment groups. Randomization will take place using the 24-hour web-based randomization system at the Fowler Kennedy Methods Centre. The computer will provide the caller with a group allocation to usual care or to the pressure management and mobility program.

Group 1: Usual Care: Subjects who are randomized to usual care will be encouraged to implement the standard wound care protocol that is consistent with the National (CAWC)and Provincial (RNAO) best practice guidelines for the treatment of pressures ulcers. This wound care program will be customized to subject's needs based on the results of the assessment performed by the wound care specialist. It will address medical, psychological, and nutritional factors interfering with wound healing and optimize the wound environment. A registered dietitian will review blood values associated with nutritional status and make recommendations for dietary changes. Wherever possible, implementation of this wound care program will be coordinated with the subjects' current health care team and appropriate referrals to home care agencies or specialists will be initiated where needed. Subjects assigned to this group will continue their current level of activity (bed rest). For the purpose of this study we have defined bed rest as a significant reduction in patient's normal activity level that involves more than 12 hours per day in bed. Any equipment or services will be obtained through the usual provider agencies and documented as part of the associated wait times. All study subjects who volunteer to participate in this screening process will receive a written report that summarizes the findings of these assessments. Included in this report will be an explanation of factors that interfere with healing and recommendations of how to modify home or wound environment to promote wound closure and limit current and future problems with skin integrity. Provided the study subject is in agreement, we will relay this information to health care professionals and administrators involved in the subject's circle of care.

Group 2: Individualized, Community-based, Pressure management and Mobility program: Subjects allocated to this group will be provided with the same customized wound care program as the usual care group and a pressure management and mobility program that is customized to the individual's needs. This program will be based on an in depth home environmental assessment(s) performed by a registered Occupational (OT) and/or Physical Therapist (PT) trained as part of the research study and will be implemented within one month of randomization.

Pressure Management program: A qualified OT or PT will examine the subject on all in-use surfaces including bed, toilet/commode, and shower chair, conduct a detailed wheelchair assessment including pressure mapping technology (X3 Pressure Mapping System, (Xsensor Technology Corporation, Calgary, Canada) and observe all transfers on and off all surfaces to identify sources of friction and shear, and any strength or balance deficits. The subject will be asked to record their activity level by completing a diary to record daily activities over a three day period including all surfaces used, duration on each surface and the number and type of transfers completed throughout the day. From this detailed 1-2 hour home assessment, the OT/PT apprentice will identify what equipment and services are required to manage pressure, improve mobility, and reduce friction and shear. Through collaboration with sponsoring company's (Waverly Glen, Shoppers Home Health, and The Roho Group). This program might include rental or purchase and installation of necessary equipment or supplies, modification of existing equipment, and follow up to provide required re-adjustments.

Mobility Program: We will contract services of a qualified Physical Therapist to assess strength, balance, range of motion, and functional independence with transfers and other ADLs. The subject will be asked to perform activities to classify their current level of functional independence using the FIM motor scale (FIM). Based on the results of this assessment she/he will develop a mobility program to optimize functional independence and improve strength and balance required for safe and effective transfers and bed mobility including educating the individual and their caregivers how to move with minimal injury to their skin. Depending on the complexity of the mobility program, delivery of this customized mobility program may involve training of the existing, community-based Personal Support Workers (PSW)s or other aids to assist with transfers, supervise strengthening and balance exercises on a regular basis.

Training of "OT/PT Apprentices" using Distance education methods: technologies A distance education model will be used to build knowledge, skills and behaviours about pressure management and rehabilitation of motor function that is needed in community based therapists - called "OT/PT Apprentices". Two therapists (OT and PT) per site will be selected and trained to implement an individualized pressure management program for people with SCI who are living in the community. They will first attend a 2 day workshop provided by L Norton and P Houghton. Information learned in this session will be reinforced using a preceptorship/mentorship model together with hands-on experience with subjects enrolled in the research study. This will begin with joint home visits with Norton and/or Houghton who will directly supervise their assessments. Subsequently, the OT/PT apprentices will perform home assessments independently and relay their findings (pressure map, room dimensions, video clips of subject transfers) electronically. Norton and Houghton will also be available by mobile phone should any questions arise during the assessments. Computer based distance learning technology (WebCT) will be used to access key articles & resources, and participate in asynchronous and synchronous discussion groups between instructors (Houghton & Norton) and Apprentices (n=4 OT or PTs). This form of eductation is know to will help foster clinical reasoning skills22-24 needed to problem solve many of the roadblocks that are anticipated with program implementation. This education program will be modified and improved throughout the study in accordance with therapist feedback and needs as identified and will inform our sixth and seventh objective.

Data & Statistical Analysis Primary Objective 1 - Wound Healing: We will calculate the percentage reduction in wound surface area for each subject by subtracting the initial wound surface area from the surface area measured at the primary endpoint - 5 months post randomization -following 3 months of the pressure management and mobility program (intervention group) or bed rest (usual care group). We will calculate the mean percentage reduction in wound surface by treatment group and determine whether the difference between groups is statistically significant using a t-test. Further, we will use an analysis of co-variance (where baseline wound surface area is entered as the covariate, wound surface area at 5 months is the dependent variable and treatment group is the independent variable) to determine whether there is statistically significant difference in the healing of pressure ulcers in individuals who receive the pressure management and mobility program compared to a similar group on bed rest, while controlling for the baseline surface area.

Objective 2 - Motor Function and Quality of Life: Similar to the analysis described above, we will use an analysis of co-variance (where the baseline measurement is entered as the covariate, the post-randomization (5 months) measure is the dependent variable and treatment group is the independent variable) to determine whether there is statistically significant difference in the quality of life (SF-12, Cardiff Wound Impact Questionnaire) in individuals who receive the pressure management and mobility program compared to a similar group on bed rest, while controlling for the baseline score. We will produce a plot to express the change in quality of life and function by time and assess whether the trajectory of change is different by group using a repeated measures analysis of covariance. As this is a pilot study, we expect to be underpowered to make statistical conclusions regarding the size of the treatment effect with confidence. However, if an important between-groups difference (20% of the minimally important difference (MID)) is contained within the 95% confidence intervals around the mean difference between groups, we will conclude that a larger study is warranted. We will provide the proportion of individuals in each group who achieve their goals as laid out in the COPM at baseline, calculate the odds of obtaining desired goals in the pressure management/mobility program compared to usual care and assess whether the difference in proportions is significant using a Fisher's Exact Test. As this is a pilot study, the study will be underpowered to confidently examine the strength of the association between motivation, caregiver burden and compliance on between-group differences. Thus, we will conduct an exploratory analysis using univariate regression methods to provide a preliminary estimate of the magnitude of the association so that we can formulate informed a priori hypotheses about the relationships between outcomes and multiple potential predictor variables that we will have sufficient power to test formally as part of the full study.

Objective 3 - Secondary Complications We will report the proportion of patients who experience adverse events by group. Adverse events will be considered any of those conditions known to commonly occur with bed rest.

Objective 4 - Cost Effectiveness: We will conduct an economic analysis to compare usual care with a pressure management/mobility program in terms of incremental cost per quality-adjusted life-year (QALY) gained from the Ministry of Health and societal perspective. The time horizon of the economic evaluation will be 8 months. To determine the 8 month direct and indirect costs associated with each alternative, resource utilization, productivity losses, informal care and out of pocket expenditures collected at baseline and at months 2, 5, and 8 will be valued using public and private sources (e.g. Ontario Schedule of Benefits for Physician Services, manufacturers). In order to calculate QALYs, utilities derived from the EQ-5D questionnaire will be weighted by time spent in health states. Regression analyses will be used in calculating QALYs to adjust for any potential differences in baseline utility values between the 2 groups.

Objective 5 Subject Recruitment: To inform our fifth objective, we will report the number of eligible patients from each source and calculate the proportion of eligible patients who are willing to participate in the study.

Objectives 6 and 7 Experiences: We will review diaries of subjects, caregivers, and therapists to optimize and streamline delivery of this program. Utilization of the methods centre as a remote, web-based, data management system will be informed by feedback from research personnel. The distance education program will be modified and improved throughout the study in accordance with "OT/PT apprentices" suggestions and needs.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-80 yrs) with a spinal cord injury (SCI) resulting in quadriplegia or paraplegia
* Stage II-IV pressure ulcer located anywhere on the body that is likely to heal over the 6 month study period.
* Requires a wheelchair for locomotion
* Able to travel to local wound centre to undergo detailed wound and medical assessment that includes blood analysis and wound culture.
* Provides consent to access relevant medical records.
* Able to adhere with study protocol, pressure management and mobility program, wound care protocol, and evaluation procedures for 8 month study period.

Exclusion Criteria:

* Unable to achieve adequate pressure relief using available resources provided by research study.
* Stage IV deep pressure sore +/- osteomyelitis that requires surgical closure.
* Medically unstable or has or any other medical condition that would prevent the individual from sitting in wheelchair for at least 2 hours (e.g. Orthostatic hypotension).
* Has a limited life expectancy that is not sufficient to complete the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Wound healing: We will measure changes in wound size and appearance using acetate tracings with Visatrak system, digital photography, and the Photographic wound assessment tool (PWAT). | monthly to 8 months post intervention

SECONDARY OUTCOMES:
Cost Effectiveness | monthly to 8 months post intervention
Quality of Life (SF-12 and Cardiff Wound Impact Questionnaire) | monthly to 8 months post intervention
Motor Performance (Canadian Occupational Performance Measure (COPM)), | monthly to 8 months post intervention
Secondary complications | monthly to 8 months post intervention
Caregiver Burden | monthly to 8 months post intervention
Compliance (diary) | monthly to 8 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Houghton, BScPT, PhD, Principal Investigator — Western University, Canada; Linda Norton, OT (Reg), Principal Investigator — Shoppers Home Health Care
Locations (2):
- Canada (2):
  - University of Western Ontario, London, Ontario
  - Women's College Hospital & Mississauga Dermatology Clinic, Toronto & Mississauga, Ontario